CLINICAL TRIAL: NCT02061085
Title: A Phase IIa Prospective, Multicenter, Open and Not Controlled of the Efficacy and Tolerability on the First Line Treatment With Eribulin as a Unic Agent on Patients With HER2 Negative Metastatic Breast Cancer Previously Treated With Taxanes
Brief Title: Monotherapy With Eribulin In Her2 Negative Metastatic Breast Cancer as a First Line Treatment
Acronym: MERIBEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-SW-H-02; 2012-004463-41 (EudraCT Number)
Record Dates: First submitted 2014-01-10; First posted 2014-02-12 (Estimated); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Breast Neoplasm; Metastasis
Keywords: Breast Neoplasm Metastasis; Receptor,HER-2; Eribulin; Furans, ketones; Antimitotic agent
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Ketosis | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- monotherapy treatment with Eribulin (Experimental): Eribulin Dosage: 1.4 mg/m2 Route of administration: IV bolus Schedule of cycle: D1 and D8 every 21 days
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin

SUMMARY:
Multicentre, prospective, non-controlled phase II clinical trial to evaluate the efficacy and tolerability of first line single agent Eribulin in patients with HER2-negative metastatic breast carcinoma (MBC) previously exposed to taxanes for early stage.

The primary objective of the study is to determine the median time to progression achieved with Eribulin. Other secondary objectives will be; overall response rate, clinical benefit rate, time to treatment progression, duration of response and toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic breast cancer HER2 negative, stage IIIb/IV
* Previous history of early disease (stage I-IIIb), surgically resected and treated with standard chemotherapy for at least 12 weeks at which included a taxane or ixabepilone
* Patients must have progressed in the 36 months after treatment with taxanes or ixabepilone.
* Age ≥ 18 years
* Given written informed consent
* Index of Eastern Cooperative Oncology Group (ECOG) of 0 or 1
* Patients must have recovered from toxicities related with previous treatment (CTC ≥ 1)
* Measurable or evaluable disease (RECIST 1.1)
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Breast cancer patients initially diagnosed with local disease advanced or metastatic disease.
* Patients who have previously received cytotoxic therapy Hormone therapy permitted if the patients have interrupted it at least two weeks before the start of the study treatment.
* Major surgery or significant traumatic injury during the 4 weeks prior to study treatment or patients who may require major surgery during the assay.
* Brain metastases or leptomeningeal uncontrolled.
* Serious medical condition and / or not properly controlled (unstable angina, lung function severe impaired, uncontrolled diabetes, active serious infection,liver disease, HIV seropositivity, active bleeding diathesis)
* Other malignancies in the last three years, except: cervical carcinoma in situ, basal cell carcinoma or squamous cell skin carcinoma,that have been properly treated
* Patients who are pregnant or breastfeeding, or adults with reproductive capacity wich are not using effective contraception.
* Patients receiving chronic treatment with systemic corticosteroids or other immunosuppressive drugs (except corticosteroids with a daily dose equivalent to prednisone ≤ 20mg on a stable dose regimen one minimum of 4 weeks prior to study entry. Topical and inhaled corticosteroids are allowed
* Active alcoholism or drugs addiction documented.
* Prior history of noncompliance with medical regimens
* Patients who do not want or can not comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, MD, Principal Investigator — Valencia
Locations (11):
- Spain (11):
  - Zaragoza, Aragon
  - Palma de Mallorca, Balearic Islands
  - Las Palmas de Gran Canaria, Canary Islands
  - Salamanca, Castille and León
  - Barcelona, Catalonia
  - Badajoz, Extremadura
  - A Coruña, Galicia
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - Madrid
  - Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 53 taxane-resistant patients with HER2- locally advanced or MBC treated with Eribulin as first-line chemotherapy were enrolled between 2013 and 2015 in a total of 14 sites.
Pre-assignment Details: Patients must comply:
  MBC HER2- stage IIIb/IV. Previous early disease (I-IIIb) diagnosis, surgically resected and treated with chemotherapy 12w (must include taxane or ixabepilone).
  Must have progressed 48m after. Age ≥ 18 years. ECOG performance status 0 or 1. Measurable or evaluable disease (RECIST 1.1). Adequate bone marrow, hepatic and renal function. Life expectancy ≥ 3m.
Period: Overall Study
Arm/Group | Monotherapy Treatment With Eribulin
Started | 53
Completed | 45
Not Completed | 8
Not completed — Adverse Event | 8

BASELINE CHARACTERISTICS:
Groups:
- Monotherapy Treatment With Eribulin: Eribulin Dosage: 1.4 mg/m2. Route of administration: IV bolus. Schedule of cycle: D1 and D8 every 21 days.
Arm/Group | Monotherapy Treatment With Eribulin
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 16
Age, Continuous [Median (Full Range); unit: years] | 47 [23 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0
Region of Enrollment [Number; unit: participants]
  Spain | 49
  Portugal | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0)
Time Frame: Through study completion, up to 27 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Monotherapy Treatment With Eribulin
Number analyzed (Participants) | 53
months | 4.1 [3.2 to 6.6]

2. Secondary Outcome: Duration of Response
Description: Duration of response
Time Frame: Through study completion, up to 27 months
Measure: Median (Full Range); unit: months
Arm/Group | Monotherapy Treatment With Eribulin
Number analyzed (Participants) | 53
months | 4.5 [2.1 to 20.9]

3. Secondary Outcome: Clinical Benefit Rate
Time Frame: Through study completion, up to 27 months
Measure: Count of Participants; unit: Participants
Groups:
- Monotherapy Treatment With Eribulin: Eribulin Dosage: 1.4 mg/m2 Route of administration: IV bolus Schedule of cycle: D1 and D8 every 21 days
  Eribulin
Arm/Group | Monotherapy Treatment With Eribulin
Number analyzed (Participants) | 53
Participants | 14

4. Secondary Outcome: Progression Free Survival
Time Frame: Through study completion, up to 27 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Monotherapy Treatment With Eribulin
Number analyzed (Participants) | 53
Months | 4.1 [3.2 to 6.6]

ADVERSE EVENTS:
Time Frame: Through study completion, up to 27 months
Arm/Group | Monotherapy Treatment With Eribulin
All-Cause Mortality (participants affected / at risk) | 22/53
Serious Adverse Events (participants affected / at risk) | 11/53
Other Adverse Events (participants affected / at risk) | 39/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monotherapy Treatment With Eribulin (N=53)
Pleural effusion (Vascular disorders) | 1 (3)
Pulmonar embolism (Vascular disorders) | 1 (3)
Cerebrovascular accident (Vascular disorders) | 1 (3)
Pulmonary tromboembolism (Vascular disorders) | 1 (2)
Cephalea (General disorders) | 1 (2)
Anxiety (General disorders) | 1 (1)
Parcial hepatoctomy (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (5)
Mucositis management (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pyelonephritis right (Renal and urinary disorders) | 1 (1)
Pyelonephritis acute (Renal and urinary disorders) | 1 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (2) — L1 fracture
Klebsiella test positive (Infections and infestations) | 1 (2)
Subcutaneous infection (Skin and subcutaneous tissue disorders) | 1 (6) — Left parascapular area
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monotherapy Treatment With Eribulin (N=53)
Neuropathy peripheral (Nervous system disorders) | 10 (10)
Dry mouth (General disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 14 (14)
Constipation (Gastrointestinal disorders) | 10 (10)
Anorexia and bulimia syndrome (Gastrointestinal disorders) | 10 (10)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (18)
Asthenia (Musculoskeletal and connective tissue disorders) | 7 (7)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No